CLINICAL TRIAL: NCT01169233
Title: Operational Evaluation of a Photic Countermeasure to Improve Alertness, Performance, and Mood During Nightshift Work on a 105-day Simulated Human Exploration Mission to Mars
Acronym: Mars 105
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Institute of Biomedical Problems (Unknown); University of Pennsylvania (Other); National Space Biomedical Research Institute (Other)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-001304; HFP00002
Record Dates: First submitted 2010-01-12; First posted 2010-07-26 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Sleep; Alertness; Fatigue
Keywords: Sleep; Alertness; fatigue; performance; spaceflight; isolation; light; Sleep , alertness and performance during a simulated spaceflight mission
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shorter Wavelength (green) (Other)
  Interventions: Device: Bright Light Box
- Intermediate Wavelength (white w/ green filter) (Other)
  Interventions: Device: Bright Light Box
- Longer Wavelength (red) (Other): Placebo
  Interventions: Device: Bright Light Box

INTERVENTIONS:
Device: Bright Light Box — Increased lighting used during night shifts to prevent sleepiness.

SUMMARY:
The success of human expedition missions critically depend on the ability of the crew to be alert and maintain high levels of cognitive function while operating complex, technical equipment. Optimal human health, performance and safety during space flight requires sufficient sleep and synchrony between the circadian pacemaker-which regulates the timing of sleep, endocrine function, alertness and performance-and the timing of the imposed sleep-wake schedule.

Crewmembers of the 105-day simulation study will be required to work one night shift every sixth night. This schedule will likely result in sleep loss and circadian misalignment, especially when lighting conditions are similar to those that crewmembers experience during spaceflight. External mission controllers will work 24-hour shifts, also resulting in both sleep loss and circadian misalignment.

It has been well documented in laboratory and field studies that both working the night shift and working extended duration shifts result in decrement alertness, performance and mood. In addition to the negative effects that night shift work has on alertness, performance and mood, shift work causes significant short and long-term health problems. Shift workers, particularly night shift workers who invert their normal sleep/wake schedule, suffer for several reasons. First, their endogenous circadian rhythms and the imposed sleep/work schedule are typically out of phase. This is similar to the experience of jet lag. However, while environment cues (e.g., sunrise, sunset, the timing of meals and sleep) enable travelers to adapt quickly to a new time zone, crewmembers in the 105-day simulation will be unable to do so because they will only spend one night of every five working. When working the night shift, the timing of meals, work, and sleep will therefore be out of phase with the normal entrained phase of the circadian timing system. Ingestion of meals at an inappropriate circadian phase results in impaired metabolism, likely underlying the gastrointestinal and metabolic problems experienced by shift workers. Second, this circadian misalignment leads to a substantial loss of sleep efficiency during the (daytime) sleep period, independent of, and in addition to, environmental obstacles to sleep (e.g., noise, light, other crewmembers). Third, misalignment of circadian phase coupled with sleep loss will each result in deterioration of alertness and impairment of performance during the night. Since these adverse effects are particularly acute on the first night of work, the plan for crewmembers on the Mars 105 mission to work the midnight shift every sixth night will subject them repeatedly to the performance impairments associated with acute circadian misalignment and acute sleep deprivation.

Lighting Countermeasure. Our group at the Harvard Medical School has successfully developed and tested effective photic countermeasures to alleviate circadian misalignment and improve alertness, performance and mood in night shift workers. The most effective countermeasure to circadian alignment is appropriately-timed and sufficiently intense light. Light also acutely improves alertness, performance and mood. Most recently it has been reported that short wavelength light has been shown to be most effective for both resetting circadian rhythms and acutely improving performance during night work via antecedent suppression of the soporific hormone melatonin.

These photic countermeasures have been tested in individual subjects living in laboratory simulations (Countermeasures readiness level/Technology readiness level 7; Evaluation with human subjects in controlled laboratory simulating operational spaceflight environment). The next critical step is to evaluate our countermeasures in an operational simulation of space flight that includes study of the interaction among crew members in a high fidelity simulation (Countermeasures readiness level/Technology readiness level 8; Validation with human subjects in actual operational spaceflight to demonstrate efficacy and operational feasibility).

Adequate sleep and circadian alignment are critical to maintaining the health and performance of expedition mission crewmembers. Testing of the developed lighting countermeasure in a high fidelity operational environment imitating the conditions of a future expedition mission (e.g., to Mars) is critical to ensure countermeasure readiness and to reduce the risk of human performance errors due to factors related to circadian disruption, sleep loss and fatigue. Development and testing of this photic countermeasure for mission controllers working 24-hour shifts will further ensure the success of the future long duration expedition missions.

DETAILED DESCRIPTION:
The objective and tasks of the investigation.

The purpose of this study is to validate the efficacy and operational feasibility of a photic countermeasure to improve alertness and performance during night shift work occurring during a simulated expedition mission. We propose to address the following specific aims:

Specific Aim 1. Evaluate the feasibility of monitoring sleep and circadian neuroendocrine rhythms in a high fidelity operational simulation of a 105-day expedition mission, in preparation for such monitoring in longer duration simulations that include the 24.65-hour Martian sol.

Specific Aim 2. Test the hypothesis that sleep, alertness, performance and mood will be impaired during acute circadian misalignment associated with night shift work operations in a high fidelity operational simulation of a 105-day expedition mission;

Specific Aim 3. Test the hypothesis that alertness, performance and mood of crewmembers exposed to shorter wavelength light (with a peak wavelength between 485 to 525 nm) during the night shift in the console monitoring room will be significantly better than the alertness, performance and mood of those same crewmembers when they are exposed to intermediate wavelength light (with a peak wavelength of either 545 nm to 555 nm) or longer wavelength light (620 nm to 690 nm) during the night shift. We hypothesize that these improvements in alertness, performance and mood will be associated with suppression of the pineal hormone melatonin. Melatonin levels are expected to be lowest across the night shift during exposure to the short 485 nm-525 nm light; low for the first quartile of the night shift during exposure to the intermediate wavelength 545 nm-555 nm light; and highest during exposure to the longer wavelength 620 nm-690 nm light. This aim will permit us to evaluate the feasibility of deploying lighting countermeasures (Light Tower; Sunnex Biotechnologies Winnipeg, Manitoba, Canada; ww.Sunnexbiotech.com) in the control panel room (inside the module EU-150) to assess the effects of this wavelength of light on alertness, performance, and subsequent sleep, in preparation for deploying lighting countermeasures in longer duration simulations that include the 24.65-hour Martian sol. Subjects will be randomized to the three lighting conditions using a balanced Latin square design.

Specific aim 4. Test the hypothesis that the alertness, performance and mood of the external mission controllers will be impaired during the final third of their extended duration, 24-hour work shifts as compared with the first third of that same work shift. We anticipate that the acute total sleep deprivation and circadian misalignment associated with hours 16 through 24 of their work shift will significantly degrade their alertness, performance and mood.

Specific aim 5. Test the hypothesis that the alertness, performance and mood of external mission controllers exposed to shorter wavelength light (with a peak wavelength between 485 to 525 nm) during the final third of their extended duration work shift will be significantly better than the alertness, performance and mood of those same crewmembers when they are exposed to intermediate wavelength light (with a peak wavelength of either 545 nm to 555 nm) or longer wavelength light (620 nm to 690 nm) during the final third of their extended duration work shift.

The purpose of the proposed studies is to address five specific hypotheses aimed at validating methods to collect data to monitor performance, sleep and circadian rhythms in an operational environment. We also plan to evaluate the efficacy of a photic countermeasure designed to improve alertness, performance, mood during acute circadian misalignment during the 105-day mission in which crewmembers will be required to be on duty in the console monitoring room during the night shift every sixth night. These five hypotheses are based on the results of our preliminary data which indicate that: (a) night shift workers who invert their normal sleep/wake schedule experience sleep loss, decreased alertness and performance; (b) individual working extended duration, 24-hour shifts experience sleep loss and impaired alertness, performance and mood, especially during a critical zone of vulnerability between the 16th and 24th hours of such extended duration work shifts; (c) shorter wavelength light acutely suppresses melatonin and increases alertness, performance and mood during night work; and (d) shorter wavelength visible light is more effective than intermediate or longer wavelength light at suppressing melatonin and increasing alertness, performance and mood during the night.

ELIGIBILITY:
The Institute of Biomedical Problems (IBMP) selected the participants for the 105-day simulated spaceflight mission. All participants that were selected by the IBMP were eligible to participate in this study.

Inclusion

* Any individual chosen by the Institute of Biomedical Problems to participate in or support the space flight simulation study was eligible to participate in the study.

Exclusion

* None. Any individual chosen by the Institute of Biomedical Problems to participate in or support the space flight simulation study was eligible to participate in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
performance on variety of cognitive tasks (e.g., psychomotor vigilance task, digit symbol substitution task) | During the 105-day isolation
sleep, measured with actigraphy | During the 105-day isolation
circadian phase | During the 105-day isolation
subjective alertness | During the 105-day isolation

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, Ph.D., M.D., Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Institute of Biomedical Problems in Moscow, Moscow, Russia

REFERENCES:
- [Background] Akerstedt T. Sleepiness as a consequence of shift work. Sleep. 1988 Feb;11(1):17-34. doi: 10.1093/sleep/11.1.17. PMID 3283910
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922
- [Background] Ashkenazi IE, Reinberg AE, Motohashi Y. Interindividual differences in the flexibility of human temporal organization: pertinence to jet lag and shiftwork. Chronobiol Int. 1997 Mar;14(2):99-113. doi: 10.3109/07420529709001148. PMID 9095371
- [Background] Brown EN, Czeisler CA. The statistical analysis of circadian phase and amplitude in constant-routine core-temperature data. J Biol Rhythms. 1992 Fall;7(3):177-202. doi: 10.1177/074873049200700301. PMID 1421473
- [Background] Budnick LD, Lerman SE, Baker TL, Jones H, Czeisler CA. Sleep and alertness in a 12-hour rotating shift work environment. J Occup Med. 1994 Dec;36(12):1295-300. doi: 10.1097/00043764-199412000-00010. PMID 7884570
- [Background] Cajochen C, Munch M, Kobialka S, Krauchi K, Steiner R, Oelhafen P, Orgul S, Wirz-Justice A. High sensitivity of human melatonin, alertness, thermoregulation, and heart rate to short wavelength light. J Clin Endocrinol Metab. 2005 Mar;90(3):1311-6. doi: 10.1210/jc.2004-0957. Epub 2004 Dec 7. PMID 15585546
- [Background] Czeisler CA, Dijk DJ. Use of bright light to treat maladaptation to night shift work and circadian rhythm sleep disorders. J Sleep Res. 1995 Dec;4(S2):70-73. doi: 10.1111/j.1365-2869.1995.tb00231.x. PMID 10607216
- [Background] Czeisler CA, Walsh JK, Roth T, Hughes RJ, Wright KP, Kingsbury L, Arora S, Schwartz JR, Niebler GE, Dinges DF; U.S. Modafinil in Shift Work Sleep Disorder Study Group. Modafinil for excessive sleepiness associated with shift-work sleep disorder. N Engl J Med. 2005 Aug 4;353(5):476-86. doi: 10.1056/NEJMoa041292. PMID 16079371
- [Background] Czeisler CA and Wright Jr. KP. Influence of light on circadian rhythmicity in humans. edited by Turek FW and Zee PC. New York: Marcel Dekker, Inc., 1999, p. 149-180.
- [Background] Di Lorenzo L, De Pergola G, Zocchetti C, L'Abbate N, Basso A, Pannacciulli N, Cignarelli M, Giorgino R, Soleo L. Effect of shift work on body mass index: results of a study performed in 319 glucose-tolerant men working in a Southern Italian industry. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1353-8. doi: 10.1038/sj.ijo.0802419. PMID 14574346
- [Background] Dubbelman M, Van der Heijde GL. The shape of the aging human lens: curvature, equivalent refractive index and the lens paradox. Vision Res. 2001 Jun;41(14):1867-77. doi: 10.1016/s0042-6989(01)00057-8. PMID 11369049
- [Background] el-Hajj Fuleihan G, Klerman EB, Brown EN, Choe Y, Brown EM, Czeisler CA. The parathyroid hormone circadian rhythm is truly endogenous--a general clinical research center study. J Clin Endocrinol Metab. 1997 Jan;82(1):281-6. doi: 10.1210/jcem.82.1.3683. PMID 8989274
- [Background] Foster RG. Neurobiology: bright blue times. Nature. 2005 Feb 17;433(7027):698-9. doi: 10.1038/433698a. No abstract available. PMID 15716938
- [Background] Gais S, Plihal W, Wagner U, Born J. Early sleep triggers memory for early visual discrimination skills. Nat Neurosci. 2000 Dec;3(12):1335-9. doi: 10.1038/81881. PMID 11100156
- [Background] Gold DR, Rogacz S, Bock N, Tosteson TD, Baum TM, Speizer FE, Czeisler CA. Rotating shift work, sleep, and accidents related to sleepiness in hospital nurses. Am J Public Health. 1992 Jul;82(7):1011-4. doi: 10.2105/ajph.82.7.1011. PMID 1609900
- [Background] Hampton SM, Morgan LM, Lawrence N, Anastasiadou T, Norris F, Deacon S, Ribeiro D, Arendt J. Postprandial hormone and metabolic responses in simulated shift work. J Endocrinol. 1996 Nov;151(2):259-67. doi: 10.1677/joe.0.1510259. PMID 8958786
- [Background] Lehrl S, Gerstmeyer K, Jacob JH, Frieling H, Henkel AW, Meyrer R, Wiltfang J, Kornhuber J, Bleich S. Blue light improves cognitive performance. J Neural Transm (Vienna). 2007;114(4):457-60. doi: 10.1007/s00702-006-0621-4. Epub 2007 Jan 25. PMID 17245536
- [Background] Lockley SW, Brainard GC, Czeisler CA. High sensitivity of the human circadian melatonin rhythm to resetting by short wavelength light. J Clin Endocrinol Metab. 2003 Sep;88(9):4502-5. doi: 10.1210/jc.2003-030570. PMID 12970330
- [Background] Lockley SW, Evans EE, Scheer FA, Brainard GC, Czeisler CA, Aeschbach D. Short-wavelength sensitivity for the direct effects of light on alertness, vigilance, and the waking electroencephalogram in humans. Sleep. 2006 Feb;29(2):161-8. PMID 16494083
- [Background] Lockley SW, Skene DJ, Arendt J, Tabandeh H, Bird AC, Defrance R. Relationship between melatonin rhythms and visual loss in the blind. J Clin Endocrinol Metab. 1997 Nov;82(11):3763-70. doi: 10.1210/jcem.82.11.4355. PMID 9360538
- [Background] Lund J, Arendt J, Hampton SM, English J, Morgan LM. Postprandial hormone and metabolic responses amongst shift workers in Antarctica. J Endocrinol. 2001 Dec;171(3):557-64. doi: 10.1677/joe.0.1710557. PMID 11739022
- [Background] Munch M, Kobialka S, Steiner R, Oelhafen P, Wirz-Justice A, Cajochen C. Wavelength-dependent effects of evening light exposure on sleep architecture and sleep EEG power density in men. Am J Physiol Regul Integr Comp Physiol. 2006 May;290(5):R1421-8. doi: 10.1152/ajpregu.00478.2005. Epub 2006 Jan 26. PMID 16439671
- [Background] Revell VL, Arendt J, Fogg LF, Skene DJ. Alerting effects of light are sensitive to very short wavelengths. Neurosci Lett. 2006 May 15;399(1-2):96-100. doi: 10.1016/j.neulet.2006.01.032. Epub 2006 Feb 21. PMID 16490309
- [Background] Ribeiro DC, Hampton SM, Morgan L, Deacon S, Arendt J. Altered postprandial hormone and metabolic responses in a simulated shift work environment. J Endocrinol. 1998 Sep;158(3):305-10. doi: 10.1677/joe.0.1580305. PMID 9846159
- [Background] Sack RL, Auckley D, Auger RR, Carskadon MA, Wright KP Jr, Vitiello MV, Zhdanova IV; American Academy of Sleep Medicine. Circadian rhythm sleep disorders: part I, basic principles, shift work and jet lag disorders. An American Academy of Sleep Medicine review. Sleep. 2007 Nov;30(11):1460-83. doi: 10.1093/sleep/30.11.1460. PMID 18041480
- [Background] Samel A, Wegmann HM. Bright light: a countermeasure for jet lag? Chronobiol Int. 1997 Mar;14(2):173-83. doi: 10.3109/07420529709001154. PMID 9095377
- [Background] Santhi N, Horowitz TS, Duffy JF, Czeisler CA. Acute sleep deprivation and circadian misalignment associated with transition onto the first night of work impairs visual selective attention. PLoS One. 2007 Nov 28;2(11):e1233. doi: 10.1371/journal.pone.0001233. PMID 18043740
- [Background] The National Uniform Crime Reporting (UCR) Program. Fact sheet for law enforcement officers killed and assaulted, 2002. 2003. [Report]
- [Background] Vener KJ, Szabo S, Moore JG. The effect of shift work on gastrointestinal (GI) function: a review. Chronobiologia. 1989 Oct-Dec;16(4):421-39. PMID 2697524
- [Background] Waterhouse J, Minors D, Redfern P. Some comments on the measurement of circadian rhythms after time-zone transitions and during night work. Chronobiol Int. 1997 Mar;14(2):125-32. doi: 10.3109/07420529709001150. PMID 9095373
- [Background] Wright KP Jr, Badia P, Myers BL, Plenzler SC. Combination of bright light and caffeine as a countermeasure for impaired alertness and performance during extended sleep deprivation. J Sleep Res. 1997 Mar;6(1):26-35. doi: 10.1046/j.1365-2869.1997.00022.x. PMID 9125696
- [Background] Wright KP Jr, Badia P, Myers BL, Plenzler SC, Hakel M. Caffeine and light effects on nighttime melatonin and temperature levels in sleep-deprived humans. Brain Res. 1997 Jan 30;747(1):78-84. doi: 10.1016/s0006-8993(96)01268-1. PMID 9042530
- [Background] Wright KP Jr, Czeisler CA. Absence of circadian phase resetting in response to bright light behind the knees. Science. 2002 Jul 26;297(5581):571. doi: 10.1126/science.1071697. No abstract available. PMID 12142528
- [Background] Wright KP Jr, Hughes RJ, Kronauer RE, Dijk DJ, Czeisler CA. Intrinsic near-24-h pacemaker period determines limits of circadian entrainment to a weak synchronizer in humans. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):14027-32. doi: 10.1073/pnas.201530198. PMID 11717461
- [Background] Wright KP Jr, Hull JT, Czeisler CA. Relationship between alertness, performance, and body temperature in humans. Am J Physiol Regul Integr Comp Physiol. 2002 Dec;283(6):R1370-7. doi: 10.1152/ajpregu.00205.2002. Epub 2002 Aug 15. PMID 12388468
- [Background] Wright KP Jr, Hull JT, Hughes RJ, Ronda JM, Czeisler CA. Sleep and wakefulness out of phase with internal biological time impairs learning in humans. J Cogn Neurosci. 2006 Apr;18(4):508-21. doi: 10.1162/jocn.2006.18.4.508. PMID 16768357
- [Background] Wright KP Jr, Myers BL, Plenzler SC, Drake CL, Badia P. Acute effects of bright light and caffeine on nighttime melatonin and temperature levels in women taking and not taking oral contraceptives. Brain Res. 2000 Aug 11;873(2):310-7. doi: 10.1016/s0006-8993(00)02557-9. PMID 10930561
- See also: Division of Sleep Medicine — http://sleep.med.harvard.edu
- See also: National Space Biomedical Research Institute — http://www.nsbri.org/